CLINICAL TRIAL: NCT02806687
Title: Phase 2 Gene Therapy Trial of Locally Advanced Pancreatic Adenocarcinoma Using Intratumoral Injection of CYL-02 in Combination With Gemcitabine
Brief Title: Effect of Intratumoral Injection of Gene Therapy for Locally Advanced Pancreatic Cancer
Acronym: THERGAP-02
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Collaborators: BIOTHERAPY department of the clinical center of investigation- CIC 1436, Toulouse (Unknown); InvivoGen Therapeutics (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC31/13/7046; 2016-000572-20 (EudraCT Number)
Record Dates: First submitted 2016-06-09; First posted 2016-06-21 (Estimated); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Pancreatic Adenocarcinoma
Keywords: Locally advanced pancreatic adenocarcinoma; gene therapy; gemcitabine; chemosensitization
MeSH Terms: interventions — Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gene Therapy product CYL-02 (Experimental): Two EUS-guided intratumor injections of CYL-02 at one month interval plus Gemcitabine (3 weeks/month) during two months followed by four months Gemcitabine alone (3 weeks/month) or until progression.
  Interventions: Drug: Gene Therapy product CYL-02; Drug: Gemcitabine
- Standard of care (Active Comparator): Gemcitabine alone 3 weeks/month during 6 months (or until progression).
  Interventions: Drug: Gemcitabine

INTERVENTIONS:
Drug: Gene Therapy product CYL-02 — Gene Therapy product CYL 02 = = plasmid DNA encoding SST2 + DCK::UMK genes pre-complexed to linear polyethylenimine.
  Intratumoral injection of the gene therapy product CYL-02 (2,5 ml within the primary tumor under endoscopic ultrasound guidance an under propofol anaesthesia). The intratumoral injection of CYL-02 is followed by three IV infusions of Gemcitabine (1000 mg/m2) at 48 hours and then every week. A second Intratumoral injection of the gene therapy product CYL-02 is performed at a same dosage and volume, 30 days after the first administration followed by three infusions of gemcitabine (1000 mg/m2) according the same rhythm (48 hours and every week) and dose. Patients have infusion of Gemcitabine 3 weeks/month during 6 months (or until progression).
  Other Names: CYL-02
  Arms: Gene Therapy product CYL-02
Drug: Gemcitabine — Gemcitabine alone 3 weeks/month during 6 months (or until progression).

SUMMARY:
Pancreatic ductal adenocarcinoma (PDAC) is the fifth leading cause of cancer-related death in Western countries, and its incidence has increased over the last 40 years. Curative surgery to manage PDAC is possible in only a fraction of patients; indeed, a vast majority (85%) of patients is diagnosed with locally advanced tumors and/or metastases because they lack specific symptoms and early markers for this disease. For these patients, palliative armamentarium consists of conventional chemotherapeutic agents such as Gemcitabine and, more recently, FOLFIRINOX, which offer marginal survival benefits. Consequently, the prognosis for PDAC is still very poor and there is great need for new treatments that can change this poor outcome. In this context, the investigators have devised, in the past few years, a highly innovative approach based on therapeutic gene transfer, which does not rely on a specific genetic and/or cellular background to inhibit PDAC tumor growth. the investigators found that SSTR2 and DCK::UMK gene transfer demonstrated complementary therapeutic effects to inhibit tumor progression and dissemination, and reduced tumor burden, respectively. On the basis of these promising preclinical data, the investigators conducted past three years the first clinical study of non-viral vector-mediated therapeutic gene delivery, guided by endoscopy (EUS), and combined with standard Gemcitabine therapy in patients with locally advanced and metastatic PDAC. The phase 1 demonstrated that the gene-therapy product CYL-02 is expressed in PDAC tumors (with long-lasting expression within tumor tissues), is distributed within the bloodstream in some extent, when combined with Gemcitabine it can inhibit primary-tumor progression and dissemination. Our results tend to demonstrate therapeutic efficacy, especially in patients with locally advanced tumors. Based on these encouraging results, the investigators propose that patients with locally advanced PDAC at the time of diagnosis may clinically benefit from this approach.

This phase II study is designed to compare the efficacy of intra-tumoral gene delivery of CYL-02 plus Gemcitabine treatment or Gemcitabine alone in patient with locally advanced PDAC.

DETAILED DESCRIPTION:
Pancreatic adenocarcinoma is the fifth leading cause of cancer related deaths in Western countries. The sole curative treatment is surgical resection. Unfortunately, curative surgery is possible in only 10 to 15 % of cases. In a palliative way, the remaining patients can be treated with chemotherapy in locally advanced (Gemcitabine) or metastatic (FOLFIRINOX) tumors. These treatments ameliorate some clinical parameters but modestly the median survival. There is an urgent need in novel treatment and gene therapy is one of these innovative approaches. The investigators demonstrated that SST2 gene (that codes for somatostatin receptor subtype 2) when transferred in pancreatic experimental tumours significantly decreases tumor progression and exerts an anti-metastatic effect. SST2 gene transfer also induced a local bystander effect due to antiproliferative, pro-apoptotic and anti-angiogenic actions. SST2 gene transfer also sensitizes pancreatic tumors to the therapeutic effect of Gemcitabine. In order to improve this chemosensitization the investigators added the DCK::UMK gene, which is a fusion between two cDNAs each coding enzymes that are critical for Gemcitabine intracellular metabolism. Effect of DCK::UMK gene transfer in combination of Gemcitabine treatment dramatically reduced the size of primary tumours in experimental models of pancreatic cancer. Finally, combining SST2 and DCK::UMK gene transfer using a single expression plasmid intratumorally injected, the investigators obtained a significant "regression" of experimental primary pancreatic tumors (Patent Cayla-INSERM 2010). In collaboration with Invivogen company, this proof of concept led us to set up a pilot Phase I clinical trial of gene therapy in unresectable pancreatic cancer patients.

For this phase I gene therapy trial (THERGAP-01NCT01274455 Dec. 2010 - Sept. 2012), the investigators produced a gene therapy product (CYL-02) in GMP grade (plasmid encoding for SST2 and DCK::UMK genes complexed to a non-viral synthetic vector PolyEthyleneImine 22 kDa). The protocol was based on two Endoscopic Ultrasound (EUS)-guided direct intratumoral injections (at one month interval) of increasing doses of DNA (125 to 1000 µg) followed by Gemcitabine infusions within 2 months. After inclusion of 22 unresectable pancreatic cancer patients the investigators demonstrated the excellent feasibility of this protocol whatever the localization of the tumor and previous treatment. No serious adverse events directly imputable to the experimental product occurred. There was no major diffusion of CYL-02 in blood (none in urine) while transgene was detected and expressed in tumour tissues in a dose-dependent manner at one month post-injection (maximum at dose 1000µg - DNA + mRNA). Primary tumor was reduced in size at one month and remained stable at 2 months with no metastatic progression in the subgroup of locally advanced patients in whom median progression-free survival and overall survival were respectively of 6.4 and 12.6 months.

These results tend to demonstrate a therapeutic effect and lead to this randomized open multicenter phase 2 trial comparing the therapeutic effect of the association "intratumoral delivery of the gene therapy product CYL-02 plus gemcitabine" versus "gemcitabine alone" in patients with locally advanced non metastatic unresectable/untreated patients.

The primary objective is to compare the effect of each modality of treatment on the progression free survival. The secondary objectives are to compare the effect on overall survival, to evaluate the antitumor response, Quality of Life local and general tolerance.

For the 6 french centers the investigators plan to include 100 patients (18 months for inclusion, 12 months for duration of the trial for each patient) with proven locally advanced non metastatic untreated pancreatic adenocarcinoma, 50 patients in each Arm: Arm A: two EUS-guided injections of CYL-02 (dose 1000 µg) at one month interval in combination of Gemcitabine infusion 1000 mg/m2 every week within two months followed by 4 months (or until progression) of Gemcitabine (same dose and rhythm); Arm B: Gemcitabine alone 1000 mg/m2 within 6 months (or until progression). In each Arm patients will be subjected to clinical and imaging follow up after 6 months including or not other treatments. CYL-02 compound will be produced and supply by DBI/Eurofins and financed by Invivogen company.

This clinical trial will be accompanied by an independent monitoring committee, which will review safety data and provide recommendations to the Sponsor regarding the safety of subjects, the conduct of the study and potential premature termination.

Evaluation will be made upon clinical symptoms, signs of tumor progression, EUS in Arm A (at one month), CT-Scan, at 2, 4, 6, 9 and 12 months (ARM A and B, RECIST 1.1 criteria). Quality of Life every month (EORTC QLC-C30 questionnaire), local and general tolerance and Pharmacokinetics of CYL-02 will be also assessed.

The dose of 1000 µg will be used and corresponds to the maximal dose tested during the phase 1b (Thergap-1). This dose demonstrated a long lasting expression within tumor, a good antitumor effect and a good tolerance (buscail et al, mol her 2015).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven local advanced pancreatic adenocarcinoma patients,
* Non metastatic locally advanced non resectable CP assessed after multidisciplinary staff* and/or surgery,
* Patient without metastasis,
* No previous antitumor treatment or pancreatic resection,
* OMS status ≤ 2,
* Measurable tumor according RECIST criteria v 1.1,
* Patient that give their informed consent,
* Patient older than 18 years of age,
* Patients no contraindication of general anaesthesia,
* Patient with primary pancreatic tumour accessible to EUS (no digestive stenosis or stomach resection).

(*: at least oncologist, radiologist, digestive surgeon and gastroenterologist)

Exclusion Criteria:

* Patients with metastatic pancreatic tumors disease,
* Contraindication of Gemcitabine infusion,
* Non-measurable primary tumour (less than 2 cm in size),
* Borderline tumour according,
* Tumour eligible to a possible neo-adjuvant treatment by radio-chemotherapy or chemotherapy (after multidisciplinary staff*),
* Contraindication to EUS-guided fine needle aspiration biopsy (coagulation disorders),
* Patient in exclusion period or participating in another clinical research protocol,
* Patient that cannot understand or read the information form / consent or is not being able to take the decision to participate to the study,
* Pregnant woman, or of childbearing potential not using contraception,
* Patient under judicial protection, guardianship or curatorship,
* Patient with cystic tumor or pancreatic pseudocyst,
* Patient bearing solid tumors other than adenocarcinoma of the pancreas (endocrine tumor, metastasis),
* Granulocytopenia: granulocytes <1000/mm3,
* Thrombocytopenia: platelet count <100 000/mm3,
* Patient not effectively treated for malignant jaundice (biliary stent or bypass) if present at diagnosis.

(*: at least oncologist, radiologist, digestive surgeon and gastroenterologist)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2017-01-30 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | From date to randomization until the date of first documented progression or date of death, whichever came first, assessed up to 12 months.
  Progression free-survival (PFS) is defined as the time interval between the date of the beginning of the treatment (Arm A: first injection of CYL-02; Arm B: first injection of Gemcitabine) and the date of local or regional progression or metastases progression or occurrence of distant metastases (including liver or non-liver metastases) or occurrence of 2nd pancreatic cancer or death (all causes), whichever occurs first. Patients alive and free of all these events will be censored at the last follow-up. Other events will be ignored (EJC 2014 Bonnetain et al).

SECONDARY OUTCOMES:
Overall survival | Up to 1 year
  Overall survival will be calculate from the date of the beginning of the treatment (Arm A: first injection of CYL-02; Arm B: first injection of Gemcitabine) until the date of death.
Tumor response | Difference between baseline and months 1, 2, 4, 6 and 12 months.
  Tumor response rates will be determined by post-therapy EUS for patients from Arm A (maximal diameter of primary tumor at 1 months versus baseline) and CT scans (Thoraco-abdominal CT - RECIST criteria 1.1 at 2, 4, 6 months versus baseline) for all patients. The overall rates for objective response (complete plus partial responses) and stable disease (no progression within 3 months) will be also considered.
Quality of life change | Difference between baseline and month 12.
  Score of Quality Of Life according to the EORTC QLQ-C30
Biological tumoral marker | Difference between baseline and month 12
  Dosage of CA 19-9 levels
Incidence of treatment-emergent adverse events | Up to 12 months
  Adverse Events, Serious Adverse Events
Biodistribution | Month 1
  Only for patient from Toulouse center: quantification of the transgene by qPCR in blood sample and tumor biopsy before and after transgene injection.
Peak plasma concentration (Cmax) | Month 1
  Only for patient from Toulouse center: quantification of the transgene by qPCR in blood sample and tumor biopsy before and after transgene injection.

CONTACTS AND LOCATIONS:
Overall Officials: Louis Buscail, MD PhD, Principal Investigator — University Hospital, Toulouse
Locations (7):
- France (7):
  - APHP Hôpital Beaujon, Clichy
  - Hôpital privé Jean Mermoz, Lyon
  - Institut Paoli Calmettes, Marseille
  - CHU de Marseille Hôpital Nord, Marseille
  - Institut régional du Cancer, Montpellier
  - Rangueil Hospital, Toulouse
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No